CLINICAL TRIAL: NCT03490695
Title: Uptake of Task-Strengthening Strategy for Hypertension Control Within Community Health Planning Services in Ghana: A Mixed Method Study.
Brief Title: Uptake of Task-Strengthening for Blood Pressure Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kintampo Health Research Centre, Ghana (Other)
Collaborators: NYU Langone Health (Other); Kwame Nkrumah University of Science and Technology (Other); St. Louis University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Kwaku Poku Asante, Director, Kintampo Health Research Centre, Ghana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 7U01HL138638-04 (NIH); 7U01HL138638-04 (NIH)
Record Dates: First submitted 2018-01-30; First posted 2018-04-06 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Hypertension; High Blood Pressure; Cardiovascular Diseases
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: For the first 12-month of the study, the intervention will not be implemented as this is a stepped-wedged design. During this time period, primary outcome (adoption ratings) and secondary outcome (Systolic BP) data will be collected at the CHPS Zones following TASSH training and the PFOs will provide support to their assigned CHPS zones to prepare to implement the TASSH protocol.
  Each CHPS zones will then be randomly assigned to one of the two intervention arms: Group A will receive the Practice Facilitation Strategy at 12 months and Group B will initially serve as a Usual Care comparison group. Group B will then receive Practice Facilitation beginning 24 months into the trial, as this is a stepped wedge design. Sustainability for groups A and B will be assessed one year after the end of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Practice Facilitation Group A (Experimental): After the first 12 months of usual care (No Practice Facilitation), group A will begin to receive the Practice Facilitation (PF) Strategy at the CHPS compounds in addition to Ghana's National Health insurance and the World Health Organization (WHO) CVD Risk Assessment package.
  Interventions: Other: Practice Facilitation; Other: Usual Care
- Practice Facilitation Group B (Experimental): Group B will receive Usual Care (no PF) between 12-24 months which includes Ghana's National Health Insurance, behavioral counseling and referral to care through the usual care system.
  After 24 months into the trial, Group B will then receive Practice Facilitation strategy in addition to Ghana's National Health insurance and the World Health Organization (WHO) CVD Risk Assessment package for a duration of another 12 months, as this is a stepped wedge design.
  During this 12 months period, practice facilitation will end in the Group A arm.
  Interventions: Other: Practice Facilitation; Other: Usual Care

INTERVENTIONS:
Other: Practice Facilitation — Community health nurses trained in implementing the evidence-based TASSH protocol will be employed as Practice Outreach Facilitators (POF) to train the CHPS community health officers to deliver TASSH. The POFs will be required to complete an intensive 12-week training course focused on adoption of TASSH protocol to identify patients at risk for uncontrolled HTN, initiate behavioral lifestyle counseling, and Refer patients to the community health centers for drug therapy. Over the course of 12 months, the POFs will provide support to their assigned CHPS zones to implement TASSH as part of routine patient care.The POFs will also work with CHPS directors to review current work flow and develop a plan of action for TASSH uptake at the CHPS zones.
Other: Usual Care — Provide Ghana's National Health Insurance, behavioral counseling and referral for care through the usual care system for 12 months.

SUMMARY:
Uptake of a community-based evidence-supported interventions for hypertension control in Ghana are urgently needed to address the cardiovascular disease epidemic and resulting illness, deaths, and societal costs. This study will evaluate the effect of Practice Facilitation on the uptake and maintenance of the evidence-based task-shifting strategies for hypertension control (TASSH) protocol across 70 Community-based Health Planning and Services (CHPS) zones delivered by trained community health officers.

Findings from this study will provide policy makers and other stakeholders the "how to do it" empirical literature on the uptake of evidence-based interventions in Ghana, which may be applicable to other low-income countries.

DETAILED DESCRIPTION:
Ghana and other countries in sub-Saharan Africa (SSA) are experiencing an epidemic of cardiovascular diseases (CVD) propelled by rapidly increasing rates of hypertension requiring implementation of evidence-based interventions. However, persistent barriers to the uptake of evidence-based interventions in low resource settings including Ghana exist at the systems, organizational and provider levels. At the systems level, lack of leadership support and shortage of staff limit effective uptake of evidence-based hypertension interventions. At the organizational level, the organizational culture, particularly the organization's readiness or openness to change may influence the use of evidence-based hypertension interventions. At the provider-level, implementation climate, lack of training, the culture of individual practices, and provider's knowledge, self-efficacy and attitude towards the evidence-based intervention limits uptake and sustainability of evidence-based interventions. The ubiquity of CHPS zones in Ghana, and their growing involvement with implementing healthcare in every community, with outreach to every doorstep, presents a unique opportunity to evaluate the effectiveness and impact of scaling up evidence-based task-shifting strategies for hypertension (TASSH) control for adults in community settings. Using a mixed methods (quantitative-qualitative) design, the investigators will evaluate practice facilitation (PF) in 70 CHPS compounds utilizing the TASSH program.

The specific aims are as follows: (1) to identify practice capacity for the adoption of TASSH at CHPS compounds and develop a culturally tailored PF strategy using qualitative methods; (2a) Evaluate in a stepped-wedge cluster Randomized Controlled trial (RCT), the effect of the PF strategy vs. Usual Care (UC), on the uptake of TASSH (primary outcome) across the CHPS compounds at 12 months;(2b) Compare in a stepped-wedge cluster RCT, the clinical effectiveness of the PF strategy vs. UC on systolic BP reduction (secondary outcome) among adults with uncontrolled hypertension at 12 months; (3) Evaluate the mediators of the uptake of TASSH across the CHPS zones at 12 months; and (4) Evaluate the sustainability of TASSH implementation across the participating CHPS compounds at 24 months (one year after completion of the trial). Outcomes will be measured every 12 months in all clusters. Guided by Damshroeder's Consolidated Framework for Implementation Research (CFIR) and Glasgow's Reach Effectiveness Adoption Implementation and Maintenance (RE-AIM) framework, the goal of this project is to improve the uptake of evidence-based task-shifting strategies for hypertension control (TASSH) in CHPS zones in Ghana. This proposal is a collaboration between the Kwame Nkrumah University of Science and Technology, Kintampo Health Research Center, New York University (NYU) School of Medicine and Saint Louis University.

ELIGIBILITY:
Inclusion Criteria

* Patients registered to receive care at CHPS zone
* Adults age 40 years and older
* Have BP 140-179/90-100 mm Hg
* Able to provide informed consent

Exclusion Criteria

* Previous diagnosis of diabetes, stroke, heart failure or chronic kidney disease BP>180/100 mm Hg
* Positive urine dipstick for protein
* Pregnant
* Unable to provide informed consent
* Patients with history of stroke, heart failure, diabetes, angina, claudication, and BP>180/100 mm Hg will be referred to a specialist

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of adoption of TASSH at the CHPS zones at 12-months | 12 months
  This is a composite measure of adoption ratings to assess the degree to which the three essential elements of the TASSH protocol (identification and screening of patients for hypertension; proportion of patients who received lifestyle counseling by the Community Health Officers (CHOs); and proportion of hypertension (HTN) patients referred for initiation of drug treatment at the CHPS zones) are adopted

SECONDARY OUTCOMES:
Systolic BP reduction at 12 months (pre- and post-intervention) | 12 months
  Change in systolic BP from baseline to 12 months
Mediators of TASSH uptake at CHPS zones at 12 months | 12 months
  Systems,organizational, and provider-level variables influencing TASSH uptake
TASSH sustainability across the participating CHPS zones one year after PF intervention ends as measured by the maintenance of TASSH adoption ratings | 12 months
  Maintenance of PF intervention effects one year after trial completion evident through sustained adoption ratings

CONTACTS AND LOCATIONS:
Overall Officials: Gbenga Ogedegbe, MD, Principal Investigator — NYU Langone Health; Kwaku Poku Asante, PhD, Principal Investigator — Kintampo Health Research Centre, Ghana; Juliet Iwelunmor, PhD, Principal Investigator — St. Louis University; Jacob Plange-Rhule, MD, Principal Investigator — Kwame Nkrumah University of Science and Technology; Kweku Bedu-Addo, PhD, Principal Investigator — Kwame Nkrumah University of Science and Technology
Locations (1):
- Kintampo Health Research Centre, Kintampo, Ghana

IPD SHARING:
Plan to Share IPD: No
Aggregate deidentified data will be shared with other researchers

REFERENCES:
- [Derived] Asante KP, Iwelunmor J, Apusiga K, Gyamfi J, Nyame S, Adjei KGA, Aifah A, Adjei K, Onakomaiya D, Chaplin WF, Ogedegbe G, Plange-Rhule J. Uptake of Task-Strengthening Strategy for Hypertension (TASSH) control within Community-Based Health Planning Services in Ghana: study protocol for a cluster randomized controlled trial. Trials. 2020 Oct 2;21(1):825. doi: 10.1186/s13063-020-04667-7. PMID 33008455